CLINICAL TRIAL: NCT07162870
Title: Idiopathic Pulmonary Fibrosis Cohort Studies of Chinese Medicine
Brief Title: Idiopathic Pulmonary Fibrosis Cohort of TCM
Status: Not yet recruiting | Type: Observational
Sponsor: Henan University of Traditional Chinese Medicine (Other)
Collaborators: The First Affiliated Hospital of Henan University of Traditional Chinese Medicine (Other); China-Japan Friendship Hospital (Other); The First Affiliated Hospital of Zhengzhou University (Other); Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Sponsor
Other Study IDs: Cohort of IPF
Record Dates: First submitted 2025-06-29; First posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-08

CONDITIONS: Idiopathic Pulmonary Fibrosis (IPF)
Keywords: Idiopathic Pulmonary Fibrosis; TCM; Cohort
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — Medicine, Chinese Traditional

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood,Tongue coating
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Traditional Chinese Medicine cohort: IPF subjects who have continuously used traditional Chinese medicine for standardized treatment for 3 months or more within 1 year, or have accumulated treatment time for 6 months or more, are classified into the traditional Chinese medicine cohort.
  Interventions: Drug: Traditional Chinese medicine (TCM)
- Non-Traditional Chinese Medicine cohort: Other IPF patients who do not meet the inclusion criteria for traditional Chinese medicine cohort, are classified into the non-traditional Chinese medicine cohort.
  Interventions: Drug: Non-traditional Chinese medicine (non-TCM)

INTERVENTIONS:
Drug: Traditional Chinese medicine (TCM) — Regulated use of Chinese medicine treatment protocols is included as an exposure factor. Exposure is defined as taking the medication continuously for more than 3 months per year, or intermittently for more than 6 months per year. According to the standardised use of TCM protocols, the group is divided into an exposed group (TCM cohort) and an unexposed group (non-TCM cohort).
  Groups: Traditional Chinese Medicine cohort
Drug: Non-traditional Chinese medicine (non-TCM) — All intervention measures that do not meet the criteria for TCM exposure are regarded as non-TCM exposure.
  Groups: Non-Traditional Chinese Medicine cohort

SUMMARY:
This study, based on past registration records, evaluates the clinical efficacy of traditional Chinese medicine in treating IPF in the real world, identifies advantageous populations and clinical targets, and provides references for precision traditional Chinese medicine treatment.

DETAILED DESCRIPTION:
This study is based on a previously established registry of interstitial lung disease, with traditional Chinese medicine treatment as the exposure factor. A total of at least 1000 IPF patients will be continuously enrolled and followed up for 2 years; it will further observe the pattern of syndromes, disease characteristics, and their interrelationships during disease development, and evaluate the clinical efficacy of traditional Chinese medicine in treating IPF using indicators such as annual acute exacerbation rate and clinical symptoms. Based on the differences in efficacy indicators, it will identify the advantageous population, clarify the clinical efficacy advantage targets, and provide a basis for precision treatment with traditional Chinese medicine.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with IPF;
2. Age ≥ 40 years old;
3. Voluntary participation in this study,And sign the informed consent form.

Exclusion Criteria:

1. Patients with confusion, dementia, consciousness disorders, and various mental illnesses;
2. Patients who are unable to take care of themselves and have been bedridden for a long time.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Idiopathic pulmonary fibrosis (IPF) is a special type of idiopathic interstitial pneumonia, which is mainly manifested by irritating dry cough and progressive dyspnea.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-09-05 (Estimated); Primary Completion 2028-10-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Annual acute exacerbation rate | Up to week 104
  The annual acute exacerbation rate will be calculated in each group at the end of the trial.

SECONDARY OUTCOMES:
Progression-Free Survival(PFS） | Evaluate the PFS at weeks 13, 26, 39, 52, 65, 78, 91, and 104.
  According to "Idiopathic Pulmonary Fibrosis in Adults (Update) and Progressive Pulmonary Fibrosis: An Official Clinical Practice Guideline of the ATS/ERS/JRS/ALAT ": The time from enrollment to the first meeting of disease progression (at least two of respiratory symptoms, physiological evidence and radiological evidence).
All-cause mortality rate | Up to week 104.
  The all-cause mortality rate will be calculated in each group at the end of the trial.
Lung transplantation rate | Up to week 104.
  The lung transplantation will be calculated in each cohort at the end of the trial.
The Traditional Chinese Medicine(TCM) Syndromes | Evaluate the TCM s]yndromes at baseline and at weeks 13, 26, 39, 52, 65, 78, 91, and 104.
  Evaluating TCM syndromes by collecting patients' symptoms, signs, tongue and pulse information.
Clinical symptoms and Signs | Evaluate the clinical symptoms and signs up at baseline and at weeks 13, 26, 39, 52, 65, 78, 91, and 104.
  Clinical symptoms and Signs will be evaluated through a scale. The scale includes coughing, expectoration, chest tightness, shortness of breath, wheezin. The Clinical Symptom Rating Scale includes 6 items: cough, expectoration, chest tightness, shortness of breath, wheezing, and cyanosis. Each item has a score of 0-3, totaling 18 points. The higher the score, the worse he patient's condition.
Forced vital capacity (FVC) | Evaluate the FVC at baseline and at weeks 26, 52, 78 and 104.
  FVC will be applied to assess pulmonary function.
FVC as the percentage of the predicted value (FVC%) | Evaluate the FVC% at baseline and at weeks 26, 52, 78 and 104.
  FVC% will be applied to assess pulmonary function.
Diffusing capacity of the lungs for carbon monoxide (DLCO) | Evaluate the DLCO at baseline and at weeks 26, 52, 78 and 104.
  DLCO will be applied to assess pulmonary function.
DLCO as the percentage of the predicted value (DLCO%) | Evaluate the DLCO% at baseline and at weeks 26, 52, 78 and 104.
  DLCO% will be applied to assess pulmonary function.
6 Six Minute Walk Distance(6MWD) | Evaluate the 6MWD at baseline and at weeks 13, 26, 39, 52, 65, 78, 91, and 104.
  The 6MWD will be applied to evaluate the exercise capacity. The higher values indicate the better exercise capacity.
The 30 - second sit - to - stand test(30s STS) | Evaluate the 30s STS at baseline and at weeks 13, 26, 39, 52, 65, 78, 91, and 104.
  The 30 second sitting and standing test will be used to evaluate lower limb strenath and cardiopulmonary function.
A Tool to Assess Quality of life (ATAQ-IPF) total scores | Evaluate the ATAQ-IPF total scores at baseline and at weeks 13, 26, 39, 52, 65, 78, 91, and 104.
  ATAQ-IPF is currently a specialized scale for evaluating the quality of life, consisting of 13 dimensions and 74 items, with each item scoring 1-5 points. The higher the score, the worse the quality of life.
St. George's respiratory questionnaire (SGRQ) total scores | Evaluate the SGRQ total scores at baseline and at weeks 13, 26, 39, 52, 65, 78, 91, and 104.
  SGRQ is a scale used to evaluate the quality of life of patients, which includes three dimensions: symptoms, mobility, and the impact of disease on daily life, with a total of 50 items. The total score range of SGRQ is usually between 0 and 100, with higher scores leading to poorer quality of life.
Dyspnea | Evaluate the mMRC total scores at baseline and at weeks 13, 26, 39, 52, 65, 78, 91, and 104.
  Dyspnea will be assessed by 22.modified Medical Research Council(mMRC) scores. A score of 0-4 will be given according to the degree of immediate dyspnea. A higher score indicates a worse condition.
C-reactive protein (CRP) | Evaluate the CRP level at baseline and at weeks 26, 52, 78 and 104.
  The CRP level will be detected by ELISA technology.
Krebs Von den Lungen-6(KL-6) | Evaluate the KL-6 level at baseline and at weeks 26, 52, 78 and 104.
  The KL-6 level will be detected by ELISA technology.
The pulmonary artery systolic pressure (PASP) | Evaluate the PASP at baseline and at weeks 26, 52, 78 and 104.
  The PASP will be measured byechocardiogram.
The diameter of the pulmonary artery | Evaluate the diameter of the pulmonary artery at baseline and at weeks 26, 52, 78 and 104.
  The diameter of the pulmonary artery will be measured byechocardiogram.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Henan University of Chinese Medicine, Zhengzhou, Henan, China